CLINICAL TRIAL: NCT06868095
Title: Multi-Center Retrospective Study to Evaluate the Impact of Sarcopenia in Patients with Early-Onset Colorectal Cancer: Incidence Risk Factor or Negative Prognosis Predictor?
Brief Title: Multi-Center Study Protocol: Impact of Sarcopenia in Early-Onset Colorectal Cancer.
Acronym: ISoPECC
Status: Enrolling by invitation | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Other Study IDs: ISoPECC Study
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Early Onset Colorectal Cancer; Sarcopenia; Prognostic Factors; Overall Survival; Disease-free Survival
MeSH Terms: conditions — Colorectal Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group: Patients < 50 years with diagnosis of colorectal cancer and with diagnosis of sarcopenia and CT-based assessment of skeletal muscle mass
  Interventions: Other: Surgical resection
- Control group: patients <50 years who had a CT- scan for suspected appendicitis or any other abdominal surgical urgency

INTERVENTIONS:
Other: Surgical resection — Histologically confirmed EOCRC
  Groups: Case group

SUMMARY:
Sarcopenia's role in early-onset colorectal cancer (EOCRC), a subtype increasingly diagnosed in individuals under 50 years, has not yet been investigated according to recent literature.

Understanding the prevalence and prognostic impact of sarcopenia in EOCRC could inform tailored therapeutic approaches and improve patient outcomes.

DETAILED DESCRIPTION:
As reported by the GLOBOCAN study, EOCRC occurs in individuals younger than 50 years old. According to the GLOBOCAN estimates, there were 188,069 new cases of EOCRC, with an Age Standardized Incidence Rate (ASRs) of 2.9 per 100,000 person-years worldwide. Recent evidence suggested an increasing incidence rate for EOCRC in different populations, with greater changes in both developed and developing countries. Despite the declining trend in the incidence of CRC in the total population of the developed countries, the incidence rates for EOCRC were increasing both in the developed and developing world. Sarcopenia's role in early-onset colorectal cancer (EOCRC), a subtype increasingly diagnosed in individuals under 50 years, remains underexplored.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed EOCRC
* Emergency room access for suspected surgical pathology
* Age: 18-49 years at diagnosis.
* Available baseline CT or MRI scans for sarcopenia assessment

Exclusion Criteria:

* Presence of comorbidity conditions severely affecting muscle mass unrelated to cancer (e.g., neuromuscular disorders).
* Inadequate follow-up data or loss to follow-up
* No past oncological history

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients younger than 50 years old who underwent colorectal cancer resection, with histologically confirmed colorectal cancer (Histologically confirmed EOCRC) and with available baseline CT or MRI scans for sarcopenia assessment
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Impact of sarcopenia on the incidence of EOCRC | Patients operated from 2000 to 2024 with at least 3 years follow-up
  Evaluation of sarcopenia on the incidence of early-onset colorectal cancer

SECONDARY OUTCOMES:
Overall survival in EOCRC patients | Patients operated from 2000 to 2024 with at least 3 years follow-up
  Assessing the overall survival in patients with diagnosis of early-onset colorectal cancer
Disease-free survival in EOCRC patients | Patients operated from 2000 to 2024 with at least 3 years follow-up
  Assessing the disease-free survival in patients with diagnosis of early-onset colorectal cancer
Prevalence of sarcopenia in EOCRC across different geographic regions | Patients operated from 2000 to 2024 with at least 3 years follow-up
  Assess the prevalence of sarcopenia in patients with diagnosis of early-onset colorectal cancer according to different geographic regions, hence how different lifestyles and nutritional habits could impact the incidence of sarcopenia
Impact of sarcopenia on post-operative complications. | Patients operated from 2000 to 2024 with at least 3 years follow-up
  Investigate how sarcopenia influences post-operative complications

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weerink LBM, van der Hoorn A, van Leeuwen BL, de Bock GH. Low skeletal muscle mass and postoperative morbidity in surgical oncology: a systematic review and meta-analysis. J Cachexia Sarcopenia Muscle. 2020 Jun;11(3):636-649. doi: 10.1002/jcsm.12529. Epub 2020 Mar 3. PMID 32125769
- [Background] Peterson SJ, Mozer M. Differentiating Sarcopenia and Cachexia Among Patients With Cancer. Nutr Clin Pract. 2017 Feb;32(1):30-39. doi: 10.1177/0884533616680354. Epub 2016 Dec 15. PMID 28124947
- [Background] Aro R, Makarainen-Uhlback E, Ammala N, Rautio T, Ohtonen P, Saarnio J, Merilainen S. The impact of sarcopenia and myosteatosis on postoperative outcomes and 5-year survival in curatively operated colorectal cancer patients - A retrospective register study. Eur J Surg Oncol. 2020 Sep;46(9):1656-1662. doi: 10.1016/j.ejso.2020.03.206. Epub 2020 Mar 17. PMID 32224072
- [Background] Roshandel G, Ghasemi-Kebria F, Malekzadeh R. Colorectal Cancer: Epidemiology, Risk Factors, and Prevention. Cancers (Basel). 2024 Apr 17;16(8):1530. doi: 10.3390/cancers16081530. PMID 38672612